CLINICAL TRIAL: NCT05507437
Title: A Participant and Investigator-blinded, Randomized, Placebo-controlled Phase 2a Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of TIN816 in Patients With Sepsis-associated Acute Kidney Injury
Brief Title: Pharmacokinetics and Safety of TIN816 in Patients With Sepsis-associated Acute Kidney Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTIN816B12201; 2022-000887-23 (EudraCT Number)
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Kidney Injury Due to Sepsis
Keywords: Sepsis; acute kidney injury; intensive care; therapy
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIN816 (Experimental): Administered as an intravenous dose
  Interventions: Biological: TIN816 70 mg lyophilisate powder
- Placebo (Placebo Comparator): 0.9% sterile sodium chloride solution administered as an intravenous dose
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TIN816 70 mg lyophilisate powder — Recombinant human CD39 enzyme
  Arms: TIN816
Other: Placebo — 0.9% sterile sodium chloride solution
  Arms: Placebo

SUMMARY:
The purpose of this study was to characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profile and to evaluate the safety and tolerability of TIN816 in hospitalized adult participants in an intensive care setting with a diagnosis of sepsis-associated acute kidney injury (SA-AKI).

DETAILED DESCRIPTION:
This was a multicenter, participant and investigator-blinded, randomized, placebo-controlled study to characterize PK/PD profile and to evaluate the safety and the tolerability of TIN816. The study enrolled hospitalized adult participants with a diagnosis of sepsis and acute kidney injury (AKI). 20 participants were randomized in the study. The study consisted of a screening period (24-48 hours), a treatment period (day 1), and post-treatment period (days 2 to 90).

Screening took place during hospitalization in a intensive care unit (ICU) (or intermediate/high dependency unit (HDU care) where potential participants were undergo screening to assess the presence of sepsis and AKI. Pre-identified participants provided informed consent and went to screening assessments to determine eligibility. Potential study candidates were hospitalized patients with a diagnosis of sepsis based on Sepsis 3 criteria with suspected or confirmed infection and SOFA score ≥ 2 after excluding the renal component, and a diagnosis of AKI stage 1 or greater. At Treatment Day 1, participants who meet eligibility criteria at screening and baseline were randomized in a 3:1 ratio to treatment with TIN816 or placebo by intravenous infusion in a participant and investigator-blinded fashion.

Treatment day 1 was followed by a 90 day post-treatment period for pharmocokinetic, pharmacodynamic, safety and tolerability assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. ≥ 18 and ≤ 85 years of age.
3. Admitted to ICU or intermediate/HDU.
4. Diagnosis of sepsis according to criteria defined by The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) based on:

   Suspected or confirmed infection SOFA score of 2 or more (excluding renal component)
5. Diagnosis of AKI Stage 1 or greater per the following criterion at randomization :

An absolute increase in serum or plasma creatinine (CR) by ≥0.3 mg/dL (≥26.5 µmol/L) within 48 hours or presumed to have occurred in the previous 48 hours as compared to the reference creatinine baseline.

For hospital-acquired AKI, a stable serum creatinine obtained in the hospital prior to AKI should be used as reference baseline, otherwise, baseline serum creatinine in the following order of preference:

Median value within 3 months of the hospital admission. If not available:

Median value between 3 and 6 months prior to hospital admission. If not available:

At hospital admission.

Exclusion criteria

1. Not expected to survive for 24 hours.
2. Not expected to survive for 30 days due to medical conditions other than SA-AKI.
3. History of CKD with a documented estimated GFR <45 ml/min prior to development of AKI.
4. Receiving RRT or a decision has been made to initiate RRT within 24 hours of admission.
5. Weight is less than 40 kg or more than 125 kg .
6. Has life support limitations (eg, do not resuscitate, do not dialyze, do not intubate).
7. AKI diagnosis according to the AKI inclusion criteria for a period longer than 48 hours prior to study drug administration.
8. Presence of AKI for a period longer than 48 hours prior to study drug administration as suggested by clinical manifestations, e.g., prolonged oliguria or severe renal dysfunction (eg, serum creatinine > 4 mg/dL) on admission without a history of CKD.
9. Evidence of recovery from AKI based on the investigator's clinical judgement prior to randomization.
10. AKI is most likely attributable to causes other than sepsis such as nephrotoxic drugs (Non-steroidal anti-inflammatory drugs (NSAIDs), contrast, aminoglycosides), other medical conditions (e.g. heart failure, liver failure, acute abdominal aortic aneurysm, dissection, renal artery stenosis) or urinary obstruction.
11. Documented (biopsy proven) or suspected history of acute or sub-acute kidney diseases such as rapidly progressive glomerular nephritis (RPGN) and acute interstitial nephritis (AIN).
12. Patients who are post-nephrectomy.
13. Patients who are on dual antiplatelet therapy.
14. Patients who are thrombocytopenic at screening (Platelet count <100,000 microliter) or other high risk for bleeding in the opinion of the investigator.
15. Immunosuppressed patients:

    History of immunodeficiency diseases or known HIV test positive. Is receiving immunosuppressant treatment or is on chronic high doses (high-dose therapy exceeding 2 weeks of treatment) of steroids equivalent to prednisone/prednisolone 0.5 mg/kg/day, including solid organ transplant patients. Patients with septic shock treated with hydrocortisone (e.g., 3 × 100 mg) can be included.
16. Active hepatitis (defined as (a) abnormal liver enzymes (Alanine aminotransferase (ALT), Gamma-glutamyl transferase (GGT), ALP > 3x Upper Limit of Normal (ULN) or (b)) for active hepatitis B or C infection, a positive Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) serology or patients with advanced chronic liver disease, confirmed by a Child-Pugh score of 10-15 (Class C).
17. Acute pancreatitis with no established source of infection.
18. Active hematological malignancy (previous hematological malignancies that are not actively treated are allowable).
19. Burns requiring ICU treatment.
20. Sepsis attributed to confirmed COVID-19.
21. Use of other investigational drugs within 5 half-lives of enrollment within 30 days (e.g., small molecules) / or until the expected pharmacodynamic effect has returned to baseline (e.g., biologics), whichever is longer; or longer if required by local regulations.
22. History of hypersensitivity to the study treatment or its excipients or to drugs of similar chemical classes.
23. Any medical conditions that could significantly increase risk of participants' safety by participating in this study according to investigator's judgement.
24. Women with a positive pregnancy test, pregnancy or breast feeding.
25. Women of child-bearing potential

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Belgium (2):
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ottignies
- France (2):
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Novartis Investigative Site, Kiel, Germany
- Novartis Investigative Site, Debrecen, Hungary
- Novartis Investigative Site, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 7 investigative sites in 5 countries.
Pre-assignment Details: The study consisted of a screening period up to 48 hours.
Groups:
- TIN816: TIN816 2 mg/kg intravenous dose on Day 1.
- Placebo: Placebo intravenous dose on Day 1
Period: Overall Study
Arm/Group | TIN816 | Placebo
Started (20) | 16 | 4
Completed (15) | 12 | 3
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIN816 | Placebo | Total
Number analyzed (Participants) | 16 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.25 (12.250) | 68.0 (19.950) | 66.60 (13.484)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 13 | 3 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 3
  Not Reported | 14 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax) of TIN816
Description: Cmax is defined as the maximum (peak) observed concentration following a dose. TIN816 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). TIN816 concentrations were determined by a validated ligand binding assay with a lower limit of quantification (LLOQ) of 10 ng/mL.
Time Frame: Day 1 (Pre-dose and 2 hours), Day 2, Day 3, Day 5, Day 8, Day 14, Day 30, Day 60 and Day 90
Population: The pharmacokinetic (PK) analysis set included all participants who survived Day 7 with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received complete study drug regardless of infusion duration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | TIN816
Number analyzed (Participants) | 16
ug/mL | 40.8 (36.7)

2. Primary Outcome: Area Under Serum Concentration-time Curve From Time Zero to the Last Measurable Concentration Sampling Time (AUClast) of TIN816
Description: AUClast is the area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (tlast) of TIN816. TIN816 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). TIN816 concentrations were determined by a validated ligand binding assay with a lower limit of quantification (LLOQ) of 10 ng/mL.
Time Frame: Day 1 (Pre-dose and 2 hours), Day 2, Day 3, Day 5, Day 8, Day 14, Day 30, Day 60 and Day 90
Population: The PK analysis set included all participants who survived Day 7 with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received complete study drug regardless of infusion duration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | TIN816
Number analyzed (Participants) | 16
day*ug/mL | 99.9 (49.0)

3. Primary Outcome: Area Under the Serum Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC[0-inf]) of TIN816
Description: The AUC from time zero to infinity (mass x time x volume-1). TIN816 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). TIN816 concentrations were determined by a validated ligand binding assay with a lower limit of quantification (LLOQ) of 10 ng/mL.
Time Frame: Day 1 (Pre-dose and 2 hours), Day 2, Day 3, Day 5, Day 8, Day 14, Day 30, Day 60 and Day 90
Population: Patients in the PK analysis set with an available value for the outcome measure. The PK analysis set included all participants who survived Day 7 with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received complete study drug regardless of infusion duration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | TIN816
Number analyzed (Participants) | 13
day*ug/mL | 104 (47.7)

4. Primary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of TIN816
Description: Tmax is the time to reach maximum (peak) drug concentration after single-dose administration (time). TIN816 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). TIN816 concentrations were determined by a validated ligand binding assay with a lower limit of quantification (LLOQ) of 10 ng/mL.
Time Frame: Day 1 (Pre-dose and 2 hours), Day 2, Day 3, Day 5, Day 8, Day 14, Day 30, Day 60 and Day 90
Population: as for outcome 2
Measure: Median (Full Range); unit: Day
Arm/Group | TIN816
Number analyzed (Participants) | 16
Day | 0.0868 [0.0597 to 0.163]

5. Primary Outcome: Terminal Elimination Half-life (T1/2) of TIN816
Description: T1/2 is the elimination half-life associated with the terminal slope. TIN816 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). TIN816 concentrations were determined by a validated ligand binding assay with a lower limit of quantification (LLOQ) of 10 ng/mL.
Time Frame: Day 1 (Pre-dose and 2 hours), Day 2, Day 3, Day 5, Day 8, Day 14, Day 30, Day 60 and Day 90
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | TIN816
Number analyzed (Participants) | 13
Day | 5.70 (14.8)

6. Primary Outcome: Total Body Clearance (CL) of TIN816
Description: CL is the total body clearance of TIN816 from the serum following intravenous administration (volume x time-1). TIN816 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). TIN816 concentrations were determined by a validated ligand binding assay with a lower limit of quantification (LLOQ) of 10 ng/mL.
Time Frame: Day 1 (Pre-dose and 2 hours), Day 2, Day 3, Day 5, Day 8, Day 14, Day 30, Day 60 and Day 90
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/day/kg
Arm/Group | TIN816
Number analyzed (Participants) | 13
Liter/day/kg | 0.0189 (24.7)

7. Primary Outcome: The Apparent Volume of Distribution (Vz) of TIN816
Description: Vz is the apparent volume of distribution during terminal phase following intravenous administration. TIN816 serum concentrations were determined using the actual recorded sampling times and non-compartmental method with Phoenix WinNonlin (Version 8.3). TIN816 concentrations were determined by a validated ligand binding assay with a lower limit of quantification (LLOQ) of 10 ng/mL.
Time Frame: Day 1 (Pre-dose and 2 hours), Day 2, Day 3, Day 5, Day 8, Day 14, Day 30, Day 60 and Day 90
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/kg
Arm/Group | TIN816
Number analyzed (Participants) | 13
Liter/kg | 0.155 (31.7)

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs (any AE regardless of seriousness) and SAEs.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 90 days.
Population: The safety analysis set (SAF) included all participants who received one dose of study treatment. Participants were analyzed according to the study treatment received, where treatment received was defined as the participants took at least one dose of that study treatment regardless treatment group randomized to.
Measure: Count of Participants; unit: Participants
Arm/Group | TIN816 | Placebo
Number analyzed (Participants) | 16 | 4
Participants
  Adverse events | 14 | 4
  Serious Adverse events | 11 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 90 days.
Groups:
- All Patients: All Patients
Arm/Group | TIN816 | Placebo | All Patients
All-Cause Mortality (participants affected / at risk) | 3/16 | 0/4 | 3/20
Serious Adverse Events (participants affected / at risk) | 11/16 | 1/4 | 12/20
Other Adverse Events (participants affected / at risk) | 14/16 | 4/4 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIN816 (N=16) | Placebo (N=4) | All Patients (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 2
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 2
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Distributive shock (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIN816 (N=16) | Placebo (N=4) | All Patients (N=20)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 5
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0 | 1
Phlyctenular keratoconjunctivitis (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3
Faecaloma (Gastrointestinal disorders) | 2 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 1
Hyperthermia (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 1
Herpes simplex reactivation (Infections and infestations) | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Skin bacterial infection (Infections and infestations) | 1 | 0 | 1
Systemic candida (Infections and infestations) | 1 | 0 | 1
Urinary tract candidiasis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 1 | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 4
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Vitamin C deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 1
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1 | 1
Myoclonus (Nervous system disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 2 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Delirium (Psychiatric disorders) | 2 | 1 | 3
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 2
Haemodynamic instability (Vascular disorders) | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2
Hypotension (Vascular disorders) | 2 | 0 | 2
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT05507437/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT05507437/SAP_001.pdf